CLINICAL TRIAL: NCT06250634
Title: Esomeprazole / Vonoprazan Combined With High-dose Amoxicillin Dual Therapy for Primary Eradication of Helicobacter Pylori Infection: a Multi-center, Prospective, Open-label, Randomized Controlled Clinical Trial
Brief Title: Esomeprazole/Vonoprazan Combined With High-dose Amoxicillin Dual Therapy for Primary Eradication of Helicobacter Pylori Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: The Second People's Hospital of Huaihua (Unknown); Yueyang Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Fen Wang, Professor, The Third Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fast 21292, Fast 23359
Record Dates: First submitted 2024-01-18; First posted 2024-02-09 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Esomeprazole; Amoxicillin; Clarithromycin; 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Double group ( Esomeprazole ) (Experimental)
  Interventions: Drug: esomeprazole + amoxicillin
- Quadruple group ( Esomeprazole ) (Active Comparator)
  Interventions: Drug: esomeprazole + amoxicillin + clarithromycin + colloidal bismuth tartrate agent
- Double group ( Vonoprazan ) (Experimental)
  Interventions: Drug: Vonoprazan + amoxicillin
- Triple group (Vonoprazan ) (Active Comparator)
  Interventions: Drug: Vonoprazan + amoxicillin + clarithromycin

INTERVENTIONS:
Drug: esomeprazole + amoxicillin — esomeprazole enteric-coated tablets (AstraZeneca) 20mg four times daily and amoxicillin capsules (Hainan General Sanyang Pharmaceutical) 750mg four times daily
  Arms: Double group ( Esomeprazole )
Drug: esomeprazole + amoxicillin + clarithromycin + colloidal bismuth tartrate agent — 20mg twice daily of esomeprazole enteric-coated tablets, 1000 mg twice daily of amoxicillin capsules, 500 mg twice daily of clarithromycin sustained-release tablets (Henan Fusen Pharmaceutical) and 165 mg three times daily of colloidal bismuth tartrate capsules (Shanxi Xinbaoyuan Pharmaceutical)
  Arms: Quadruple group ( Esomeprazole )
Drug: Vonoprazan + amoxicillin — 20 mg twice daily of vonoprazan fumarate tablets (Takeda Pharmaceutical Company Limited) and 1000 mg three times daily of amoxicillin capsules (Hainan General Sanyang Pharmaceutical)
  Arms: Double group ( Vonoprazan )
Drug: Vonoprazan + amoxicillin + clarithromycin — 20 mg twice daily of vonoprazan fumarate tablets, 1000 mg twice daily of amoxicillin capsules and 500 mg twice daily of clarithromycin sustained-release tablets (Henan Fusen Pharmaceutical)
  Arms: Triple group (Vonoprazan )

SUMMARY:
This study intends to collect the clinical data of patients with Helicobacter pylori infection, and to observe and count the high-dose double therapy and the traditional quadruple / triple therapy ( i.e., esomeprazole + amoxicillin double high-dose double therapy and esomeprazole + amoxicillin + clarithromycin + colloidal bismuth tartrate traditional quadruple therapy or Vonoprazan + amoxicillin double high-dose double therapy and Vonoprazan + amoxicillin + clarithromycin triple therapy ). The eradication rate of Helicobacter pylori was compared between the two different regimens respectively, and the efficacy, safety and compliance of different regimens were compared. It provides a new reference for clinical treatment of Helicobacter pylori, and has great clinical value and significance for simplifying the anti-Helicobacter-pylori treatment plan, increasing patient compliance, and exploring efficient anti-Helicobacter-pylori therapy suitable for the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 14-90 years, no requirement for gender;
2. patients diagnosed as H. pylori infection by at least one of the following tests: carbon-13/14 urea breath test (13C/14C-UBT) or immuno-histochemical staining of biopsy specimens;
3. patients with no use of antibiotics, bismuth or Chinese traditional medicines with antibacterial effects in the previous 4 weeks of 13C/14C-UBT, and no H2 receptor antagonists, PPIs, P-CAB or other drugs affecting H .pylori activity within the previous 2 weeks of 13C/14C-UBT;
4. patients without history of receiving H. pylori eradication therapy.

Exclusion Criteria:

1. patients with serious diseases or clinical conditions that may interfere with the evaluation of the results of the study, such as severe heart, liver, lung, and renal insufficiency, low immunity, and so on;
2. patients with allergy to penicillin or any research-program-related drugs;
3. patients with mental illness and communication disorders;
4. patients in pregnancy or lactation;
5. patients with severe gastrointestinal diseases, such as gastrointestinal tumors, gastrointestinal bleeding, other organic diseases, etc.;
6. patients who were participating in other clinical trials;
7. patients who were considered inappropriate for enrollment after evaluation by the researchers.

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | pre-intervention and at least 30 days post-intervention
  carbon-13/14 urea breath test

SECONDARY OUTCOMES:
Adverse events | the 3rd, 7th, and 14th day during the intervention
Compliance | the 14th day during the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- outpatient department of gastroenterology of the Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No